CLINICAL TRIAL: NCT03601325
Title: Acute Pancreatitis: Study of Possible Etiologies and Risk Factors Affecting Outcome (Hospital Based Study)
Brief Title: Acute Pancreatitis: Study of Possible Etiologies and Risk Factors Affecting Outcome
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SMMostafa, Specialist of tropical medicine and gastroenterology, Assiut University
Other Study IDs: Acute pancreatitis
Record Dates: First submitted 2018-05-21; First posted 2018-07-26 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Pancreatitis
Keywords: pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to assess the frequency of different etiologies of acute pancreatitis in our locality & assess the effect of different risk factors on outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

-

Diagnosis of acute pancreatitis according to the following: the presence of two of the three following criteria:

* abdominal pain consistent with the disease
* serum amylase and or lipase greater than three times the upper limit of normal
* characteristic findings from abdominal imaging Contrast-enhanced computed tomographic (CECT) and or magnetic resonance imaging (MRI) of the pancreas

Exclusion Criteria:

* No exclusion criteria .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in assuit university hospital during the period of the study and diagnosed as acute pancreatitis
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
The frequency of different etiologies of AP in our locality | 1 year
  At the end of study, total number of patients of each etiology of acute pancreatitis will be calculated as (Gallstones, Alcohol, triglyceridemia, Idiopathic, ERCP,..)

SECONDARY OUTCOMES:
Outcome of the patients according to the Atlanta Classification 2012 revision | 1 year
  Effect of each risk factor on outcome as progression to mild, moderate severe and severe pancreatitis "according to the Atlanta Classification 2012 revision",
Hospital duration of stay | 1 year
  Effect of each risk factor on hospital duration of stay
Rate of transfer to ICU | 1 year
  Effect of each risk factor on rate of transfer to ICU
Mortality | 1 year
  Effect of each risk factor on mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Osman, MD, Study Director — Assiut University
Locations (1):
- Ahmed Mohammed Abu-Elfatth, Asyut, Egypt